CLINICAL TRIAL: NCT05595265
Title: Expression of Programmed Death Ligand-1 (PD-L1) in Nasopharyngeal and Hyypopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nahaweend Mohamed Hafez, demonstrator, pathology department, faculty of medicine, sohag university, Sohag University
Other Study IDs: Soh_Med_22_10_20
Record Dates: First submitted 2022-10-23; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Nasopharyngeal and Hypopharyngeal Carcinoma
MeSH Terms: conditions — Hypopharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: immunohistochemical — Immunohistochemical Evaluation: Corresponding sections of 4µm thickness from each Formalin-fixed paraffin blocks will be immunohistochemically stained by anti- PD-L1 antibody according to the recommended protocol.

SUMMARY:
Head and neck tumors comprise heterogeneous neoplasms that arise from surface epithelium of different anatomic subsites in head and neck region such as oral cavity, oropharynx, larynx and hypopharynx. Nasopharyngeal and hypopharyngeal carcinomas represent 0.26 % of all cancers in Egypt. Tobacco exposure and alcohol dependence, and infection with oncogenic viruses such as human Papilloma virus (HPV) are among the risk factors for development of these tumors. Currently, the main treatment of nasopharyngeal and hypopharyngeal carcinomas is radio-chemotherapy based in histological type, grade and stages of the tumors

Tumor infiltrating lymphocytes (TILs) are considered as cornerstone in cancer immunotherapy and as a biomarker with effectiveness predictive value. The intensity and quality of immune cells, especially lymphocytes, in tumor microenvironment are strongly related to the outcome of immune checkpoint blockade therapy .

ELIGIBILITY:
Inclusion Criteria:

* Patients with nasopharyngeal and hypopharyngeal carcinomas who underwent diagnostic biopsies.

Exclusion Criteria:

* Patients received chemotherapy or radiotherapy.
* Patients with insufficient clinical data.
* Specimens with extensive necrosis
* Tiny specimens which are insufficient for accurate diagnosis.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: - Patients with nasopharyngeal and hypopharyngeal carcinomas who underwent diagnostic biopsies.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
expression of programmed death ligand-1 (PD-L1) in nasopharyngeal and hypopharyngeal carcinoma | 12 months
  evaluate expression of PD-L1 in nasopharyngeal and hypopharyngeal carcinomas and to correlate its expression to different clinical and histopathological parameters to address its prognostic value.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Background] Mehanna H, Beech T, Nicholson T, El-Hariry I, McConkey C, Paleri V, Roberts S. Prevalence of human papillomavirus in oropharyngeal and nonoropharyngeal head and neck cancer--systematic review and meta-analysis of trends by time and region. Head Neck. 2013 May;35(5):747-55. doi: 10.1002/hed.22015. Epub 2012 Jan 20. PMID 22267298
- [Background] Willenbrink TJ, Ruiz ES, Cornejo CM, Schmults CD, Arron ST, Jambusaria-Pahlajani A. Field cancerization: Definition, epidemiology, risk factors, and outcomes. J Am Acad Dermatol. 2020 Sep;83(3):709-717. doi: 10.1016/j.jaad.2020.03.126. Epub 2020 May 7. PMID 32387665
- [Background] Paijens ST, Vledder A, de Bruyn M, Nijman HW. Tumor-infiltrating lymphocytes in the immunotherapy era. Cell Mol Immunol. 2021 Apr;18(4):842-859. doi: 10.1038/s41423-020-00565-9. Epub 2020 Nov 2. PMID 33139907